CLINICAL TRIAL: NCT07273539
Title: A Randomised, Controlled, Examiner Blind Study to Evaluate the Effect of a Sodium Bicarbonate Toothpaste on the Oral Microbiome
Brief Title: A Study to Evaluate the Effect of a Test (Sodium Bicarbonate) Toothpaste on the Oral Microbiome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 400039
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — sodium bicarbonate-based toothpaste

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Toothpaste (Experimental): Participants will be instructed to brush their teeth with the test toothpaste for at least one minute twice daily (morning and evening) for 12 weeks.
  Interventions: Drug: Sodium Bicarbonate Toothpaste
- Reference Toothpaste (Active Comparator): Participants will be instructed to brush their teeth with the reference toothpaste for at least one minute twice daily (morning and evening) for 12 weeks.
  Interventions: Drug: Sodium Fluoride Toothpaste

INTERVENTIONS:
Drug: Sodium Bicarbonate Toothpaste — A toothpaste containing sodium bicarbonate and sodium fluoride.
  Arms: Test Toothpaste
Drug: Sodium Fluoride Toothpaste — A toothpaste containing 0.315 percent (%) weight/weight (w/w) sodium fluoride; 1450 parts per million (ppm) fluoride.
  Arms: Reference Toothpaste

SUMMARY:
The aim of this 12-week clinical study is to evaluate the effect of a toothpaste containing sodium bicarbonate over time on the oral microbiome and to explore its effect in comparison to a regular fluoride toothpaste in participants with localized gingivitis.

DETAILED DESCRIPTION:
This will be a single-center, 12-week, randomized, controlled, single-blind (examiner only), two-treatment arm, parallel group design, clinical study investigating the effect of a toothpaste containing sodium bicarbonate on the oral microbiome in healthy adult participants with mild-moderate gingivitis. Approximately 55 participants (approximately 27 per group) will be randomized to ensure approximately 50 evaluable participants (approximately 25 per group) complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant's biological sex at birth was male or female.
* Participant who, at the time of screening is aged 18-65 years, inclusive.
* A participant who is willing and able to comply with scheduled visits, treatment plan and other study procedures.
* A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon oral examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* Participant with at least 20 natural, permanent teeth (excluding 3rd molars) and with at least 40 evaluable surfaces.
* A healthy participant with mild to moderate gingivitis in the opinion of the clinical examiner.

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or a Haleon employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant who has any other clinical serious or unstable conditions (example, cardiovascular diseases, diabetes, liver disorders, and kidney disorders) which could have affected study out comes and/or participant safety.
* A participant who is a pregnant female (self-reported) at screening or baseline visit or intending to become pregnant over the duration of the study or who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant unwilling or unable to comply with the Lifestyle Considerations described in this protocol (these will be added in the full protocol).
* A participant who is a current smoker or an ex-smoker (including vaper) who stopped within 6 months of Screening.
* A participant who is using smokeless forms of tobacco (example, chewing tobacco, gutkha, pan containing tobacco, nicotine-based e-cigarettes).
* A participant who is diagnosed with oral dryness or is taking any medication that in the view of the investigator is causing oral dryness.
* A participant who has a medical condition which could have directly influenced gingival bleeding.
* A participant who has a bleeding disorder that could have affected study outcomes and/or participant safety.
* A participant who has a recent history (within the last year) of alcohol or other substance abuse.
* A participant who has a severe oral condition (example, acute necrotizing ulcerative gingivitis or oral or peri-oral ulceration including herpetic lesions) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant/examiner if they participate in the study.
* Presence of a tongue or lip piercing, or any other oral feature that could interfere with the usage of a toothbrush.
* A participant using any antibiotic and/or probiotic medication within 28 days prior to screening or at any time during the study.
* Participant who has used an oral care product containing anti-bacterial (example, chlorhexidine), probiotic or other ingredient that, in the opinion of the investigator or dentally qualified designee, could affect plaque formation or gingival health within 4 weeks of Screening or between Screening and the Baseline visit.
* A participant currently taking an anti-inflammatory medication which, in the opinion of the Investigator, could affect gingival condition.
* A participant currently taking an anti-inflammatory medication which, in the opinion of the Investigator, could affect gingival condition.
* A participant currently taking a systemic medication (example, anti-inflammatory, anticoagulant, immunosuppressants) or traditional/herbal remedy which, in the opinion of the Investigator, could affect plaque/ gingival condition (example, ibuprofen, aspirin, warfarin, cyclosporin, phenytoin, calcium channel blockers).
* A participant who shows signs of periodontitis or is receiving or has received treatment for periodontal disease (including surgery) within 12 months of Screening.
* A participant who has gingivitis, which in the opinion of the investigator, is not expected to respond to treatment with an over the counter (OTC) dentifrice.
* A participant who has active caries that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they participate in the study.
* A participant who has dentures (partial or full).
* A participant who has Fixed orthodontic appliances or is undergoing active or recent (within 3 months of Screening) orthodontic treatment, which in the opinion of the investigator, could interfere with study procedures, assessments or outcomes.
* A participant who has other orthodontic devices (example, bands, fixed retainers, or removable retainers) that could, in the opinion of the investigator, interferes with study procedures, assessment or outcomes.
* A participant who has numerous restorations in a poor state of repair.
* A participant who has any dental condition (example, overcrowding) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they participate in the study.
* A participant who has had dental prophylaxis within 12 weeks of Screening.
* A participant who has had teeth bleaching within 12 weeks of Screening.
* A participant who has high levels of extrinsic stain or calculus deposits
* A participant who has previously been enrolled in this study.
* A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Bacterial Composition at Week 12 by Treatment Groups | Baseline and Week 12
  Taxonomic changes of microbial communities in plaque samples will be reported.

SECONDARY OUTCOMES:
Change From Baseline in Potential Bacterial Activity at Week 12 by Treatment Groups | Baseline and Week 12
  Potential functional capabilities of microbial communities in plaque samples will be reported in different areas of plaque.
Differences in Bacterial Composition at Week 12 (Test Toothpaste Versus (Vs) Control Toothpaste) | Week 12
  Comparison of bacterial composition in different areas of plaque will be reported.
Differences in Bacterial Composition Between Different Areas of Plaque at Week 12 | Week 12
  Comparison of bacterial composition in different areas of plaque will be reported for test and reference toothpaste.

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Sharma, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.